CLINICAL TRIAL: NCT02839720
Title: Pilot Study of the MEK1/2 Inhibitor Selumetinib (AZD6244 Hydrogen Sulfate) for Adults With Neurofibromatosis Type 1 (NF1) and Cutaneous Neurofibromas (CNF)
Brief Title: Selumetinib in Treating Patients With Neurofibromatosis Type 1 and Cutaneous Neurofibroma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01087; NCI-2016-01087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9990 (Other: University of Alabama at Birmingham Cancer Center); 9990 (Other: CTEP); P30CA013148 (NIH); NCT03105258 (obsolete NCT alias)
Record Dates: First submitted 2016-07-20; First posted 2016-07-21 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cutaneous Neurofibroma; Neurofibromatosis Type 1; Optic Nerve Glioma
MeSH Terms: conditions — Neurofibromatosis 1; Optic Nerve Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selumetinib sulfate) (Experimental): Patients receive selumetinib sulfate PO twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience a volume decrease in the target cutaneous neurofibromas may continue treatment for 12 additional cycles.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib Sulfate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate

SUMMARY:
This pilot phase II trial studies how well selumetinib works in treating patients with neurofibromatosis type 1 and cutaneous neurofibromas. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine if selumetinib sulfate (selumetinib) can result in shrinkage of cutaneous neurofibromas.

SECONDARY OBJECTIVE:

I. Assess the effect of selumetinib on target inhibition in cutaneous neurofibroma(s) excised prior treatment and on treatment with selumetinib for analysis of percent inhibition of phosphorylated ERK (pERK), and changes in phosphorylated AKT (pAKT).

EXPLORATORY OBJECTIVES:

I. Assess the effect of selumetinib on the development on new cutaneous neurofibromas while on treatment with selumetinib.

II. Assess the effect of selumetinib on target inhibition in cutaneous neurofibroma(s) excised prior treatment and on treatment with selumetinib for analysis of the tumor kinome.

III. Assess the effect of selumetinib skin related morbidity and pain using the Skindex, the Global Impression of Change Scale and Numeric Rating Scale, all of which are patient reported outcome measures.

IV. Quantify the development of new cutaneous neurofibromas on treatment with selumetinib.

V. Detailed pathologic analysis of cutaneous neurofibromas pretreatment and on treatment with selumetinib for changes in cell composition (including macrophage and mast cell infiltration).

VI. Investigate alterations that correlate with cutaneous neurofibroma (cNF) response to selumetinib treatment with pilot genomic, deoxyribonucleic acid (DNA) methylation, and transcriptomic studies.

OUTLINE:

Patients receive selumetinib sulfate orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience a volume decrease in the target cutaneous neurofibromas may continue treatment for 12 additional cycles.

After completion of study treatment, patients are followed up every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients be >= 18 years old at the time of enrollment and must have a documented germline neurofibromatosis 1 (NF1) mutation in a Clinical Laboratory Improvement Act (CLIA) certified laboratory or a diagnosis of NF1 based on clinical National Institutes of Health (NIH) consensus criteria; in addition to substantial cutaneous neurofibroma burden, at least one of the criteria below have to be present

  * Six or more cafe-au-lait macules (>= 0.5 cm in prepubertal subjects or >= 1.5 cm in post pubertal subjects)
  * Freckling in axilla or groin
  * Optic glioma
  * Two or more Lisch nodules
  * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
  * A first-degree relative with NF1
  * Histologic confirmation of tumor is not necessary in the presence of consistent clinical findings
* Patients must have substantial cutaneous neurofibroma burden causing distress to the patient by disfigurement or itching; patients must have >= 9 measurable cutaneous neurofibromas; for the purpose of this study measurability will be defined for each of the lesions selected as target lesions as a neurofibroma with a longest diameter >= 4 mm in the longest diameter
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin >= 10 g/dL (not requiring red blood cell [RBC] transfusions)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL (not requiring platelet transfusions)
* Total bilirubin =< 1.5 X upper limit of normal (ULN), with the exception of patients with Gilbert syndrome who are required to have =< 3 X ULN
* Alanine transferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 X ULN
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability of subject or legally authorized representative (LAR) to understand and the willingness to sign a written informed consent document
* Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated
* Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g. grapefruit juice or marmalade) during the study
* Since there is no standard effective chemotherapy for patients with NF1 and cutaneous neurofibromas, patients may be treated on this trial without having received prior medical therapy directed at their plexiform neurofibromas (PN)
* Since selumetinib is not expected to cause substantial myelosuppression, there will be no limit to number of prior myelosuppressive regimens previously received for NF1 related; or other tumor manifestations
* Patients who have received previous investigational agents or biologic therapy, such as tipifarnib, pirfenidone, Peg-intron, sorafenib, or other vascular endothelial growth factor (VEGFR) inhibitors are eligible for enrollment
* Growth factors that support platelet or white cell number or function must not have been administered within the past 7 days and are not permitted while on the study
* At least 6 weeks must have elapsed prior to enrollment since the patient received any prior radiation therapy, and the target cutaneous neurofibromas have to be in areas outside of a prior radiation field
* At least 4 weeks must have elapsed since receiving medical therapy directed at NF1 related tumor manifestations
* At least 4 weeks must have elapsed since any surgeries, with evidence of completed wound healing
* Patients who received prior medical therapy for a NF1 related tumor must have recovered from the acute toxic effects of all prior therapy to =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 before entering this study
* The effects of selumetinib on the developing human fetus at the recommended therapeutic dose are unknown; for this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 weeks after dosing with selumetinib ceases; women of child-bearing potential must have a negative pregnancy test prior to entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform her treating physician immediately; please note that the selumetinib manufacturer recommends that adequate contraception for male patients should be used for 12 weeks post-last dose due to sperm life cycle
* Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent from all patients, which can be accomplished using the study specific informed consent or another consent, such as the National Cancer Institute (NCI), Pediatric Oncology Branch (POB) screening protocol; studies or procedures that were performed for clinical indications (not exclusively to determine eligibility) may be used for screening or baseline values even if the studies were done before informed consent was obtained, if the patient agrees

Exclusion Criteria:

* Patients who are receiving any other investigational agents, or have received an investigational agent within the past 30 days
* May not have a NF1 related tumor such as optic pathway glioma or malignant peripheral nerve sheath tumor, which requires treatment with chemotherapy, radiation, or surgery
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements; patients with HIV who have adequate cluster of differentiation (CD)4 counts and who have no requirement for antiviral therapy will be eligible
* Pregnant or breast-feeding females are excluded due to potential risks of fetal and teratogenic adverse events of an investigational agent; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method; abstinence is an acceptable method of birth control
* Prior treatment with selumetinib or another specific MEK 1/2 inhibitor
* No supplementation with vitamin E is permitted
* Inability to swallow capsules, since capsules cannot be crushed or broken
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Strong inhibitors or inducers of hepatic microsomal isoenzymes
* While not an exclusion criterion, unless clinically indicated, patients should avoid taking other additional non-study medications that may interfere with the study medications; in particular, patients should avoid medications that are known to strong inhibitor or inducers of hepatic microsomal isoenzymes CYP1A2, CYP2C8, CYP2C9, CYP2C19, CYP3A4/5, UGT1A1, UGT1A3 and transporters BCRP and P-gp
* Known cardiac disorder, including:

  * Uncontrolled hypertension (blood pressure [BP] of >= 150/95 despite medical support/management)
  * Acute coronary syndrome within 6 months prior to starting treatment
  * Uncontrolled angina - Canadian Cardiovascular Society grade II-IV despite medical support/management
  * Heart failure New York Heart Association (NYHA) class II or above
  * Prior or current cardiomyopathy including but not limited to the following:

    * Known hypertrophic cardiomyopathy
  * Known arrhythmogenic right ventricular cardiomyopathy
  * Baseline left ventricular ejection fraction (LVEF) =< 53%
  * Previous moderate or severe impairment of left ventricular systolic function (LVEF < 40% on echocardiography or equivalent on multi-gated acquisition scan [MUGA]) even if full recovery has occurred
  * Severe valvular heart disease
  * Atrial fibrillation with a ventricular rate > 100 beats per minute (bpm) on electrocardiography (ECG) at rest
  * Fridericia's correction formula (QTcF) interval > 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) are excluded; the use of medication(s) that can prolong corrected QT (QTc) interval is prohibited while treated on this study
* Known ophthalmologic conditions, such as:

  * Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR)
  * Current or past history of retinal vein occlusion
  * Known intraocular pressure (IOP) > 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP); patients with controlled glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) may be eligible after discussion with the study chair
  * Subjects with any other significant abnormality on ophthalmic examination (performed by an ophthalmologist) should be discussed with the study chair for potential eligibility
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
* Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib
* Have had recent major surgery within a minimum of 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access
* Have any unresolved chronic toxicity with CTCAE grade >= 2, from previous anti-NF1 therapy, except for alopecia
* Clinical judgment by the investigator that the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R Korf, Principal Investigator — University of Alabama at Birmingham Cancer Center
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Derived] Gross AM, Reid OH, Baldwin LA, Cannon A, Choo-Wosoba H, Steinberg SM, Lobbous M, Wolters PL, Pichard DC, Tibery CM, Dombi E, Derdak J, Widemann BC, Korf BR. Treatment of Cutaneous Neurofibromas in Neurofibromatosis Type 1 With MEK Inhibitor Selumetinib: A Nonrandomized Clinical Trial. JAMA Dermatol. 2025 Feb 26;161(5):533-7. doi: 10.1001/jamadermatol.2024.6574. Online ahead of print. PMID 40009403
- [Derived] Church C, Fay CX, Kriukov E, Liu H, Cannon A, Baldwin LA, Crossman DK, Korf B, Wallace MR, Gross AM, Widemann BC, Kesterson RA, Baranov P, Wallis D. snRNA-seq of human cutaneous neurofibromas before and after selumetinib treatment implicates role of altered Schwann cell states, inter-cellular signaling, and extracellular matrix in treatment response. Acta Neuropathol Commun. 2024 Jun 21;12(1):102. doi: 10.1186/s40478-024-01821-z. PMID 38907342

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Selumetinib): Participants receive selumetinib capsules at a dose of 50mg by mouth (PO) twice daily (BID) every 12 hours with option to increase to 75mg PO BID after first cycle if tolerated. Treatment repeats every 28 days (1 cycle = 28 days) for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Participants who experience a volume decrease in the target cutaneous neurofibromas may continue treatment for 12 additional cycles. Volume decrease defined as a greater than or equal to 20 percent decrease in the sum of the volumes of the smaller and/or larger target cutaneous neurofibromas.
Period: Overall Study
Arm/Group | Treatment (Selumetinib)
Started | 11
Completed | 4
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Non-compliance | 2
Not completed — Intercurrent Illness | 1
Not completed — Non-compliance due to COVID-19 pandemic | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Average cutaneous neurofibroma (cNF) volume [Mean (Full Range); unit: microliters] | 159.1 [42.4 to 425.4]

OUTCOME MEASURES:

1. Primary Outcome: Median Best Response of Cutaneous Neurofibromas in Participants With at Least One Restaging Evaluation
Description: Average percent change in volume of target cutaneous neurofibromas from baseline. Cutaneous neurofibromas measured with calipers and volumes calculated by multiplying length, width and height of each target neurofibroma. At each response evaluation (baseline and then after every 4 cycles), the sum of the on-treatment volumes for the target cutaneous neurofibromas were subtracted from the pre-treatment volumes of the same tumors to arrive at an overall percentage change in target cutaneous neurofibroma size for each participant at each restaging evaluation. The average percent change that was most decreased from baseline (best response) for each participant was collected and the timepoint at which this occurred was noted. The median and range of these average percent change best responses are reported here.
Time Frame: Up to 24 cycles of treatment (1 cycle = 28 days)
Population: Includes all participants who had at least one restaging evaluation on treatment with selumetinib
Measure: Median (Full Range); unit: percent change
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 8
percent change | -28.5 [-84.9 to 24.8]

2. Secondary Outcome: Change in the Number of Cutaneous Neurofibromas
Description: At the time of each response evaluation (baseline and then after every 4 cycles), the number of cutaneous neurofibromas (cNFs) that are greater than 4mm as measured with a caliper were counted in the picture frames. We report here the change in overall number of cutaneous neurofibromas counted after 12 cycles of treatment (Number of cNFs counted after 12 cycles - Number of cNFs counted at baseline).
Time Frame: Baseline to up to 1 year
Population: Includes all participants that completed 12 cycles of selumetinib.
Measure: Median (Full Range); unit: neurofibromas
Groups:
- Treatment (Selumetinib): Participants receive selumetinib capsules at a dose of 50mg by mouth (PO) twice daily (BID) every 12 hours with option to increase to 75mg PO BID after first cycle. Treatment repeats every 28 days (1 cycle = 28 days) for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Participants who experience a volume decrease in the target cutaneous neurofibromas may continue treatment for 12 additional cycles. Volume decrease defined as a greater than or equal to 20 percent decrease in the sum of the volumes of the smaller and/or larger target cutaneous neurofibromas.
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 5
neurofibromas | -7 [-30 to 4]

3. Other Pre Specified Outcome: Changes in Skin Related Morbidity
Description: Assessed by Skindex. Global Impression of Change Scale and Numeric Rating Scale evaluations were not used in this outcome measure due to limited data set. Skindex is a dermatology survey whose scores are normalized to a 0-100 scale with higher scores indicating worse quality of life. We report here the change in overall Skindex score after 12 cycles of treatment (Score at 12 cycles - Score at Baseline).
Time Frame: Baseline to up to 1 year
Population: Only included analysis of the 5 participants who had baseline and 1 year on treatment Overall SkinDex scores available.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Treatment (Selumetinib Sulfate): Participants receive selumetinib capsules at a dose of 50mg by mouth (PO) twice daily (BID) every 12 hours with option to increase to 75mg PO BID after first cycle if tolerated. Treatment repeats every 28 days (1 cycle = 28 days) for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Participants who experience a volume decrease in the target cutaneous neurofibromas may continue treatment for 12 additional cycles. Volume decrease defined as a greater than or equal to 20 percent decrease in the sum of the volumes of the smaller and/or larger target cutaneous neurofibromas.
Arm/Group | Treatment (Selumetinib Sulfate)
Number analyzed (Participants) | 5
score on a scale | -1.72 [-15.52 to 12.07]

4. Other Pre Specified Outcome: Changes in Pathway Biomarkers Assessed by Kinome Analysis
Description: Will be tested for statistical significance using a Wilcoxon signed rank test.
Time Frame: Baseline to up to 1 year
Population: Trial was terminated due to low accrual that was exacerbated by the COVID-19 pandemic leading to limited data set for this outcome measure. Not enough samples to justify proceeding with this analysis.
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Changes in Levels of pERK and pAKT Assessed by Quantitative Enzyme-linked Immunosorbent Assay
Description: Will be correlated with tumor volume changes using Spearman rank correlation. Exploratory comparisons between patients with a tumor response and those without a response will be done using a Wilcoxon rank sum test.
Time Frame: Baseline to up to 1 year
Population: as for outcome 4
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline through study completion, a maximum of 36 cycles (approximately 3 years)
Arm/Group | Treatment (Selumetinib)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Selumetinib) (N=11)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Posterior Vitreous Detachment OD, Grade 2, Attribution = Unlikely
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) — Drug Reaction with Eosinophilia and Systemic Symptoms, Grade 3, Attribution = Possible
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unknown abdominal mass, Grade 3, Attribution = Unrelated
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) — Grade 4, Attribution = Unlikely
Hypertension (Vascular disorders) | 1 (2) — Grade 4, Attribution = Possible
Hypertension (Vascular disorders) | 1 (2) — Grade 3, Attribution = Unlikely
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Selumetinib) (N=11)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Constipation (Gastrointestinal disorders) | 2 (22) — Grade 1
Constipation (Gastrointestinal disorders) | 1 (2) — Grade 2
Diarrhea (Gastrointestinal disorders) | 4 (32) — Grade 1
Dry mouth (Gastrointestinal disorders) | 1 (15) — Grade 1
Gastrointestinal disorders - Other, specify (Dark stools) (Gastrointestinal disorders) | 1 (2) — Grade 1
Nausea (Gastrointestinal disorders) | 2 (13) — Grade 1
Nausea (Gastrointestinal disorders) | 1 (17) — Grade 2
Vomiting (Gastrointestinal disorders) | 1 (2) — Grade 1
Vomiting (Gastrointestinal disorders) | 1 (2) — Grade 2
Edema face (General disorders) | 1 (2) — Grade 1
Edema limbs (General disorders) | 3 (7) — Grade 1
Fatigue (General disorders) | 2 (40) — Grade 1
Fatigue (General disorders) | 1 (2) — Grade 2
Flu like symptoms (General disorders) | 1 (1) — Grade 1
Alanine aminotransferase increased (Infections and infestations) | 2 (7) — Grade 2
Aspartate aminotransferase increased (Infections and infestations) | 2 (29) — Grade 1
Aspartate aminotransferase increased (Infections and infestations) | 1 (10) — Grade 2
Paronychia (Infections and infestations) | 1 (13) — Grade 1
Alanine aminotransferase increased (Investigations) | 1 (17) — Grade 1
Alkaline phosphatase increased (Investigations) | 1 (10) — Grade 1
CPK increased (Investigations) | 3 (48) — Grade 1
CPK increased (Investigations) | 1 (5) — Grade 2
Lipase increased (Investigations) | 2 (13) — Grade 1
Serum amylase increased (Investigations) | 1 (8) — Grade 1
Serum amylase increased (Investigations) | 1 (2) — Grade 2
Dizziness (Nervous system disorders) | 1 (2) — Grade 1
Dysgeusia (Nervous system disorders) | 1 (15) — Grade 1
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) — Grade 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 (6) — Grade 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 (88) — Grade 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 (15) — Grade 2
Nail loss (Skin and subcutaneous tissue disorders) | 1 (3) — Grade 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 (5) — Grade 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (100) — Grade 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (41) — Grade 2
Skin and subcutaneous tissue disorders - Other, specify (Onchomycosis) (Skin and subcutaneous tissue disorders) | 2 (25) — Grade 1
Skin and subcutaneous tissue disorders - Other, specify (Skin fissures) (Skin and subcutaneous tissue disorders) | 1 (3) — Grade 1
Hypertension (Vascular disorders) | 1 (2) — Grade 1
Hypertension (Vascular disorders) | 2 (16) — Grade 2

LIMITATIONS AND CAVEATS:
Study was terminated early by CTEP due to low accrual but allowed participants who were already on study to continue to receive treatment if they were responding or had stable disease. Low accrual was exacerbated by the COVID-19 pandemic leading to a small number of subjects analyzed and with many subjects having missing data or evaluations due to an inability to travel to the study site. Due to the limited data set, we are only able to provide descriptive analyses of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT02839720/Prot_SAP_000.pdf